CLINICAL TRIAL: NCT02132429
Title: Phase I, Randomized, Double-Blind, Placebo-Controlled, Ascending Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 333 in Healthy Subjects and Migraine Subjects
Brief Title: Phase I, Double-Blind,Placebo, MAD Study to Evaluate the Safety, Tolerability, PK, and PD of AMG 333 in Healthy Subjects and Migraine Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was stopped due to an administrative decision not safety.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20130246
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Migraine
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — AMG 333

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 333 (Experimental): Subjects will receive a single oral dose of AMG 333 daily for 14 days.
  Interventions: Drug: AMG 333
- Placebo (Placebo Comparator): Subjects will receive a single oral dose of placebo daily for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 333 — Oral administration available in varying dose strength.
  Arms: AMG 333
Drug: Placebo — Placebo containing no active drug
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of multiple oral doses of AMG 333 for 14 days in healthy subjects and migraine subjects. As part of the secondary objectives, the study will characterize the pharmacokinetic (PK) profile of AMG 333 after multiple oral doses in healthy subjects and migraine subjects, as well as characterize the effect of multiple doses of AMG 333 on increases in blood pressure (BP) induced by the cold pressor test (CPT) in healthy subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, ascending multiple-dose study evaluating AMG 333 in healthy subjects and subjects with migraines. Eight healthy subjects will be enrolled in each of cohorts 1 through 5. Study subjects will be randomized such that 6 subjects will receive AMG 333 and 2 subjects will receive placebo (3:1 ratio) per cohort. Likewise, 8 migraine subjects will be enrolled in cohort 6 and randomized to receive AMG 333 or placebo (3:1 ratio). All subjects will be housed for 15 days then allowed to return home. Migraine subjects will self-administer the headache diary at least once daily during the screening and out-patient portions of the study, and site personnel will administer the headache diary during the in-house period of the study. Healthy subjects will not keep the headache diary during screening and will have the headache diary administered by site personnel at least once daily starting on day 1 through day 14, and will then self administer throughout their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects (cohorts 1 through 5) and male and female subjects with migraines (cohort 6), who are ≥ 18 and ≤ 55 years of age at the time of screening, and have no history or evidence of clinically-relevant medical disorders as determined by the investigator in consultation with the Amgen physician.

Exclusion Criteria:

* History or evidence of a clinically significant disorder, condition, or disease that in the opinion of the investigator and Amgen physician, would significantly impair pain perception (eg, history of stroke, history of neuropathy), would pose a risk to subject safety or interfere with evaluation, procedures, or study completion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent AEs | Up to 29 Days
  Treatment-emergent adverse events, including changes in vital signs, 12-lead ECGs, clinical laboratory safety tests, and physical and neurological assessments

SECONDARY OUTCOMES:
Plasma PK Parameter | Up to 29 Days
  Plasma PK parameters of AMG 333: time to maximum concentration (tmax)
Plasma PK Parameter | Up to 29 Days
  Maximum observed concentration (Cmax)
Plasma PK Parameter | Up to 29 Days
  Area Under the Concentration Time-Curve from time 0 to 24 hours postdose (AUC0-24) and Days 1 and 14
Blood Pressure response to CPT | Up to 29 Days
  Change in systolic and diastolic BP in response to the CPT in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- CRI Lifetree, Salt Lake City, Utah, United States

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com